CLINICAL TRIAL: NCT05232617
Title: The Effects of Online Rheumatological Rehabilitation Education on Readiness, Clinical Decision Making and Perceived Self-efficacy in Intern Physiotherapy Students
Brief Title: The Effects of Online Rheumatological Rehabilitation Education in Intern Physiotherapy Students
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assist. Prof., Istanbul University - Cerrahpasa
Other Study IDs: 09/12/2020-161414
Record Dates: First submitted 2021-06-17; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Learning Problem
Keywords: Learning management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatological rehabilitation training
  Interventions: Other: Rheumatological rehabilitation training

INTERVENTIONS:
Other: Rheumatological rehabilitation training — Online rheumatological rehabilitation training is planned. Online rheumatological rehabilitation training will be video-based via the Edpuzzle application and interactively via the zoom application. Online trainings are planned for 15-person intern physiotherapy student groups 4 days a week, 2 hours a day, for 4 weeks on a case-based basis. With the Edpuzzle application, videos will be prepared for 10 different rheumatological diseases. In each video, a case with rheumatic disease will be introduced, evaluations made from a physiotherapy perspective and their results will be included. Before the lesson, students will watch the video defined for them every day from the application called Edpuzzle, answer the questions and plan a disease-specific assessment and treatment program according to the directions in the video. Then, the assessment and treatment programs prepared by a group of 15 people through the zoom platform will be discussed during the lesson.

SUMMARY:
The aim of the study is to investigate the effect of online rheumatological rehabilitation training on readiness, clinical decision making and perceived self-efficacy in intern physiotherapy students. In the study, online rheumatological rehabilitation training is planned. Online rheumatological rehabilitation training will be video-based via the Edpuzzle application and interactively via the zoom application. Online trainings are planned for 15-person intern physiotherapy student groups 4 days a week, 2 hours a day, for 4 weeks on a case-based basis. In the study, readiness, clinical decision making and perceived self-efficacy levels will be evaluated in intern physiotherapy students before and after online rheumatological rehabilitation training.

ELIGIBILITY:
Inclusion Criteria:

* To be taking Rheumatological Rehabilitation internship course

Exclusion Criteria:

* To have taken the Rheumatological Rehabilitation Internship course before, but failed to complete it successfully
* Lack of internet access

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Intern physiotherapy students taking the Rheumatology Internship course at Istanbul University Cerrahpaşa Faculty of Health Sciences, Physiotherapy and Rehabilitation will be included in the study. In the 2020-2021 academic year, 60 intern physiotherapy students who took the Rheumatology Internship course will be included. Consent will be obtained from all participants with a voluntary information form on google forms.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Readiness Scale for Mobile Learning | Change from baseline to 4 weeks
  Mobile Learning Readiness Scale will be used to determine students' readiness for mobile learning. Scale, Lin et al. and Gokcearslan et al. adapted to Turkish and its validity and reliability were made. While there are 19 items in the original version of the scale, there are 17 items in the Turkish version. Scale items; "self-efficacy (items 1-2-3-4-5-6), optimism (items 7-8-9-10-11-12-13), and self-learning (items 14-15-16-17)" are grouped. The variance rate of the scale was 76.9% and the internal consistency coefficient (Cronbach alpha) was 0.95. The reliability coefficient of the scale is 0.959. The items in the scale are 7-point Likert type; degree of agreement is scored between (1) "I strongly disagree" and (7) "I strongly agree". The lowest 17 points and the highest 119 points can be obtained from the scale. The data are evaluated over the total score.

SECONDARY OUTCOMES:
Melbourne Decision-Making Scale I-II | Change from baseline to 4 weeks
  Students' clinical decision making skills Mann et al. "Melbourne Decision-Making Scale (MKVÖ) I-II" was developed to determine the self-esteem and decision-making styles of university students in decision-making. It consists of six items and a single sub-factor, and three items are scored straight and three items are scored in the opposite direction. "Correct" answer given to scoring items is made as 2 points, "Sometimes True" answer is 1 point, "Not True" answer is given 0 points. The maximum score that can be obtained from the scale is 12. High scores indicate high self-esteem in decision making. II. Part (MCDS II): It consists of 22 items and measures decision-making styles. High scores indicate the use of the relevant decision-making style. It has four sub-factors. They are Mindful Decision Making Style (6 items), Avoidant Decision Making Style (6 items), Procrastinating Decision Making Style (5 items) and Panic Decision Making Style (5 items). This scale is answered like MKVÖ I.
General Self-Efficacy Scale | Change from baseline to 4 weeks
  Students' self-efficacy levels will be evaluated with the General Self-Efficacy Scale. This scale is a measurement tool for self-assessment. The Turkish validity and reliability study of the scale was conducted by Yıldırm et al. made by. In the scale, there are five reversed items and two positive statements. The score of each question varies between 1-5. An increase in the total score indicates an increase in self-efficacy belief.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided